CLINICAL TRIAL: NCT00368667
Title: Energy Homeostasis in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK 02749 (completed)
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Body Composition; Metabolic Rate
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the potential biological predispositions that contribute to the difficulty patients with anorexia nervosa have in maintaining normal weight.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a psychiatric illness that is characterized by extreme weight loss and severe body image distortions. In this study, we are examining changes in body composition, metabolic rate, and reproductive function before and after treatment for AN. More specifically, we are testing the hypotheses that 1)Weight-restored patients with AN have elevated resting energy expenditure (REE) compared to controls, 2) Weight-restored patients with AN have a central disposition of body fat compared to controls, 3) Weight-restored patients with AN who gain the most fat centrally will have the least improvement on psychological measures, 4) Weight-restored patients with AN will have leptin levels out of proportion to body fat mass. It will also investigate the relationship between REE and leptin with respect to the return of menses.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* DSM-IV diagnosis of Anorexia Nervosa
* BMI ≤ 17.5kg/m2 (equivalent to 80% of ideal body weight)
* Medically stable
* Participation in in-patient treatment sufficient to restore patient to a BMI of at least 19kg/m2

Exclusion Criteria:

* On medication*
* Current substance abuse or dependence
* History of suicide attempt or other self-injurious behavior within the previous 6 months
* Non-removable metal on/in their body (e.g. metal pacemaker, surgical clips, metallic-ink tattoos)

Controls:

Inclusion criteria:

* No current psychiatric disorder (including eating disorder, depression, bipolar disorder, schizophrenia, substance abuse/dependence)
* No history of an eating disorder
* BMI greater than 19kg/m2 and less than 21kg/m2
* Weight stable (+/- 2kg) for the previous 6 months
* No history of excessive or repeated dieting
* No history of excessive exercise (defined as greater than 6 hours/week)
* Regular menstrual cycles

Exclusion criteria:

* On medication*
* Pregnant or lactating
* Significant medical problem
* Non-removable metal on/in their body (e.g. metal pacemaker, surgical clips, metallic-ink tattoos)

  * At the time of testing, subjects will be free of fluoxetine for 6 weeks, and free of all other medications for a minimum of 2 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2000-04; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Mayer, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, Unit 98, New York, New York, United States

REFERENCES:
- [Result] Mayer L, Walsh BT, Pierson RN Jr, Heymsfield SB, Gallagher D, Wang J, Parides MK, Leibel RL, Warren MP, Killory E, Glasofer D. Body fat redistribution after weight gain in women with anorexia nervosa. Am J Clin Nutr. 2005 Jun;81(6):1286-91. doi: 10.1093/ajcn/81.6.1286. PMID 15941877
- [Derived] Schebendach J, Mayer LE, Devlin MJ, Attia E, Walsh BT. Dietary energy density and diet variety as risk factors for relapse in anorexia nervosa: a replication. Int J Eat Disord. 2012 Jan;45(1):79-84. doi: 10.1002/eat.20922. Epub 2011 Mar 29. PMID 21448937
- [Derived] Bodell LP, Mayer LE. Percent body fat is a risk factor for relapse in anorexia nervosa: a replication study. Int J Eat Disord. 2011 Mar;44(2):118-23. doi: 10.1002/eat.20801. PMID 20127939
- [Derived] Mayer LE, Klein DA, Black E, Attia E, Shen W, Mao X, Shungu DC, Punyanita M, Gallagher D, Wang J, Heymsfield SB, Hirsch J, Ginsberg HN, Walsh BT. Adipose tissue distribution after weight restoration and weight maintenance in women with anorexia nervosa. Am J Clin Nutr. 2009 Nov;90(5):1132-7. doi: 10.3945/ajcn.2009.27820. Epub 2009 Sep 30. PMID 19793856